CLINICAL TRIAL: NCT01150955
Title: Potential Beneficial Effects of Resveratrol on Obesity, Metabolic Syndrome and Inflammation - Emphasis on Description of the Molecular Biology Underpinning the Interplay Between Calorie Restriction, SIRT1, STAT5 and the GH/IGF-I Axis
Brief Title: Potential Beneficial Effects of Resveratrol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: M-20100058
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: Resveratrol; Diabetes; SIRT1; STAT5; IGF-I; Growth hormone; NAFLD; Longevity; Substrate metabolism; Calorie restriction
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Diabetes Mellitus; Non-alcoholic Fatty Liver Disease | interventions — Resveratrol; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resveratrol (Active Comparator): Dietary supplement of resveratrol 500 mg three times a day over five weeks.
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — 500 mg three times a day for five weeks.
  Other Names: Fluxome Sciences.
  Arms: Resveratrol
Other: Placebo — Placebo (starch capsules) 500 mg three times a day for five weeks.
  Other Names: Starch
  Arms: Placebo

SUMMARY:
We want to investigate whether the food supplement resveratrol is able to counteract the detrimental effects of obesity.

DETAILED DESCRIPTION:
The aim of this study is to investigate potential metabolic effects of resveratrol in healthy but obese men. We hypothesize that resveratrol will counteract some of the detrimental effects of obesity, and as an imitator of calorie restriction will give new insight into the basic biochemical pathways underpinning human metabolism. Of special interest is the potential connection between resveratrol, calorie restriction, SIRT1, STAT5b and the GH/IGF-I axis.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2
* Otherwise healthy
* Written informed consent

Exclusion Criteria:

* Any disease
* Alcohol dependency
* Allergy to trial medication
* Present or previous malignancy
* Participation in other clinical trials within three months before randomization

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Metabolic parameters | Five weeks
  Regarding glucose, protein and fat metabolism.

SECONDARY OUTCOMES:
Pathways of substrate metabolism. | Five weeks
  Description of the biochemical pathways underpinning the interplay between calorie restriction, SIRT1, STAT5 and the GH/IGF-I axis.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jørgensen, Professor,MD, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Endocrinology, MEA, Aarhus, Denmark

REFERENCES:
- [Derived] Clasen BF, Poulsen MM, Escande C, Pedersen SB, Moller N, Chini EN, Jessen N, Jorgensen JO. Growth hormone signaling in muscle and adipose tissue of obese human subjects: associations with measures of body composition and interaction with resveratrol treatment. J Clin Endocrinol Metab. 2014 Dec;99(12):E2565-73. doi: 10.1210/jc.2014-2215. PMID 25050904
- [Derived] Poulsen MM, Vestergaard PF, Clasen BF, Radko Y, Christensen LP, Stodkilde-Jorgensen H, Moller N, Jessen N, Pedersen SB, Jorgensen JO. High-dose resveratrol supplementation in obese men: an investigator-initiated, randomized, placebo-controlled clinical trial of substrate metabolism, insulin sensitivity, and body composition. Diabetes. 2013 Apr;62(4):1186-95. doi: 10.2337/db12-0975. Epub 2012 Nov 28. PMID 23193181